CLINICAL TRIAL: NCT05522972
Title: Improving Normal and Amblyopic Vision With Video Games and Perceptual Learning
Brief Title: Establishing New Treatment Approaches for Amblyopia: Perceptual Learning and Video Games
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Roger W. Li, Associate Professor, Nova Southeastern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-344
Record Dates: First submitted 2022-08-24; First posted 2022-08-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Amblyopia
Keywords: perceptual learning; video games; visual plasticity; amblyopia treatment; pathophysiology of amblyopia; vision training; stereoacuity; strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Games (Experimental): Participants will be required to play video games for a period of time: 1-2 hrs per session, 4-5 sessions/week for ~1-6 months
  Interventions: Behavioral: Video Game Vision Training
- Perceptual learning (Experimental): Participants will be required to practice a visual discrimination task (e.g. visual acuity, position acuity, contrast sensitivity, & stereoacuity) for a period of time: 1-2 hrs per session, 4-5 sessions/week for ~1-6 months
  Interventions: Behavioral: Perceptual Learning
- Occlusion therapy (Active Comparator): Participants will be required to cover the dominant eye during the day in order to push the brain to use the fellow amblyopic eye: 1-2 hrs per session, 4-5 sessions/week for ~1-6 months
  Interventions: Behavioral: Occlusion Therapy

INTERVENTIONS:
Behavioral: Video Game Vision Training — A new approach for improving amblyopic vision using video games
  Arms: Video Games
Behavioral: Perceptual Learning — A new approach for improving amblyopic vision with perceptual learning
  Arms: Perceptual learning
Behavioral: Occlusion Therapy — Conventional treatment for amblyopia
  Arms: Occlusion therapy

SUMMARY:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. This study uses psychophysical measures to study neural plasticity in both adults and children with amblyopia.

DETAILED DESCRIPTION:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. Our previous findings (see Publications) show that the adult amblyopic brain is still plastic and malleable, suggesting that active approach is potential useful in treating amblyopia.The goal of this project is to assess the limits and mechanisms of neural plasticity in both normal and amblyopic spatial vision. This study uses psychophysical measures to study neural plasticity in both adults and children with amblyopia. Research participants will be asked to practice a visual discrimination task (perceptual learning) or to play video games with the amblyopic eye for a period of time. A range of visual functions will be monitored during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* adults and children with normal vision or amblyopia
* amblyopia: interocular VA difference of 0.1 logMAR or more

Exclusion Criteria:

* any ocular pathological conditions, nystagmus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity before and after the intervention | 9 months
  "Visual acuity", the gold standard for vision testing, will be measured. Participants will be asked to read letters on a LogMAR letter chart. The smallest letters that can be read correspond to visual acuity (e.g., Snellen acuity of 20/20, letter-stroke width = 1 minute of arc).
Change in stereoacuity before and after the intervention | 9 months
  "Stereoacuity" will be measured psychophysically using a new stereoacuity function test (1.25, 2.5, 5, 10, 15, & 20 cycles per degree) developed in our previous studies (Li et al 2016). A custom-built 4-mirror haploscope will be used to present a stereogram to each eye. Stereoacuity is the smallest stereo disparity that can be seen in binocular vision (in the unit of seconds of arc, arcsec).
  The conventional stereoacuity tests (including Randot Stereoacuity Test, Stereofly Test & Preschool Stereo Test) will also be used to measure stereoacuity. Participants will be asked to wear a pair of 3D glasses and to identify the target 3D pictures at various 3D levels. The smallest 3D disparities that can be seen correspond to stereoacuity (e.g. normal range of stereoacuity: 50 seconds of arc or better).

SECONDARY OUTCOMES:
Change in contrast sensitivity before and after the intervention | 9 months
  "Contrast sensitivity", the ability to detect low contrast / brightness, will be measured psychophysically for a range of spatial frequencies (1.25, 2.5, 5, 10, & 20 cycles per degree). Visual stimuli at different contrast levels will be displayed on a monitor screen. The smallest detectable stimulus contrast level will be measured in the unit of cd/m2.
Change in positional (or Vernier) acuity before and after the intervention | 9 months
  "Positional acuity", the ability to detect a subtle positional offset between visual stimuli, will be measured psychophysically. Visual stimuli with different amount of positional offsets will be displayed on a monitor screen. The smallest detectable stimulus offset will be measured as position acuity, in the unit of seconds of arc.

CONTACTS AND LOCATIONS:
Overall Officials: Roger W Li, OD, PhD, Principal Investigator — Nova Southeastern University College of Optometry
Locations (1):
- Nova Southeastern University College of Optometry, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li RW, Li BZ, Chat SW, Patel SS, Chung STL, Levi DM. Playing three-dimensional video games boosts stereo vision. Curr Biol. 2024 Jun 3;34(11):R524-R525. doi: 10.1016/j.cub.2024.04.032. PMID 38834021
- [Background] Leung TW, Li RW, Kee CS. Brief Adaptation to Astigmatism Reduces Meridional Anisotropy in Contrast Sensitivity. Invest Ophthalmol Vis Sci. 2023 Sep 1;64(12):4. doi: 10.1167/iovs.64.12.4. PMID 37656478
- [Background] Li RW, Levi DM. Characterizing the mechanisms of improvement for position discrimination in adult amblyopia. J Vis. 2004 Jun 1;4(6):476-87. doi: 10.1167/4.6.7. PMID 15330715
- [Background] Bahnson BJ, Anderson VE. Isotope effects on the crotonase reaction. Biochemistry. 1989 May 16;28(10):4173-81. doi: 10.1021/bi00436a008. PMID 2765479
- [Background] Li RW, Provost A, Levi DM. Extended perceptual learning results in substantial recovery of positional acuity and visual acuity in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2007 Nov;48(11):5046-51. doi: 10.1167/iovs.07-0324. PMID 17962456
- [Background] Li RW, Young KG, Hoenig P, Levi DM. Perceptual learning improves visual performance in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3161-8. doi: 10.1167/iovs.05-0286. PMID 16123415
- [Background] Li RW, Ngo CV, Levi DM. Relieving the attentional blink in the amblyopic brain with video games. Sci Rep. 2015 Feb 26;5:8483. doi: 10.1038/srep08483. PMID 25715870
- [Background] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514
- [Background] Li RW, Tran KD, Bui JK, Antonucci MM, Ngo CV, Levi DM. Improving Adult Amblyopic Vision with Stereoscopic 3-Dimensional Video Games. Ophthalmology. 2018 Oct;125(10):1660-1662. doi: 10.1016/j.ophtha.2018.04.025. Epub 2018 May 18. No abstract available. PMID 29779684
- [Background] Li RW, Tran TT, Craven AP, Leung TW, Chat SW, Levi DM. Sharpening coarse-to-fine stereo vision by perceptual learning: asymmetric transfer across the spatial frequency spectrum. R Soc Open Sci. 2016 Jan 20;3(1):150523. doi: 10.1098/rsos.150523. eCollection 2016 Jan. PMID 26909178
- [Background] Li RW, So K, Wu TH, Craven AP, Tran TT, Gustafson KM, Levi DM. Monocular blur alters the tuning characteristics of stereopsis for spatial frequency and size. R Soc Open Sci. 2016 Sep 21;3(9):160273. doi: 10.1098/rsos.160273. eCollection 2016 Sep. PMID 27703690
- [Background] Li RW, Levi DM, Klein SA. Perceptual learning improves efficiency by re-tuning the decision 'template' for position discrimination. Nat Neurosci. 2004 Feb;7(2):178-83. doi: 10.1038/nn1183. Epub 2004 Jan 18. PMID 14730311